CLINICAL TRIAL: NCT00749294
Title: Measurement of Anogenital Wart Burden, and Cost of Illnesses in Bangkok
Brief Title: Anogenital Wart Burden and Cost of Illnesses
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Prof. Punnee Pitisuttithum, Mahidol University
Other Study IDs: THALS1570
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-08

CONDITIONS: Warts
MeSH Terms: conditions — Warts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation

SUMMARY:
The study will be a prospective study of patients presenting with anogenital warts. The objective are to assess proportion of anogenital warts to the total number of sexual transmitted infection patients, to quantify direct and indirect cost of illnesses and psychological burden associated with anogenital warts and to estimate government program expenditure for the prevention and control and treatment of the STI/anogenital HPV infection.

DETAILED DESCRIPTION:
An observational study, multiple visit, 2-center study will be conducted in Rajavithi General Hospital, and Bangrak Hospital. One hundred and fifty subjects will be enrolled from both hospitals. Anogenital wart patients presented in Rajavithi General Hospital and the STI clinic at Bangrak Hospital will be recruited prospectively. All patients will be treated according to standard medical guidelines or usual care of the institutes. After the baseline assessment, the patients will have follow up visits with their physicians and will also be interviewed at the clinical sites three time approximately at day 7 (-2+7 days), month 1 (+-7 days), and month 6 (+-7 days) until they are cure. At month 6 (+-14 days), telephone assessment for the capture of any signs of disease recurrence will be done. All patients will be followed for 6 months under the same schedule.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older and has anogenital warts
* Physician confirmed clinical diagnosis of anogenital warts
* Subject is capable of understanding the study and the content of the consent form and has agreed to participate in the study by signing the informed consent
* Subject will be available for the study follow up period

Exclusion Criteria:

* Subject is unable to give informed consent
* Subject has any condition which in the opinion of the investigator might interfere with the evaluation of the study objectives such as other concurrent/active STI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with anogenital warts, conducted at Rajavithi General Hospital and Bangrak Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Punnee Pitisuttithum, M.B.,B.S., Principal Investigator — Mahidol University
Locations (1):
- Clinical Infectious Diseases Research Unit, Bangkok, Bangkok, Thailand